CLINICAL TRIAL: NCT04546074
Title: Imatinib Mesylate in Combination With Pembrolizumab in Patients With Advanced KIT-mutant Melanoma Following Progression on Standard Therapy: a Phase I/II Trial
Brief Title: Imatinib Mesylate in Combination With Pembrolizumab in Patients With Melanoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Keio University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Ohara Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Takeru Funakoshi, Assistant Professor, Keio University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N20190002
Record Dates: First submitted 2020-08-29; First posted 2020-09-11 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Melanoma
Keywords: KIT
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Pembrolizumab and Imatinib mesylate

INTERVENTIONS:
Drug: Pembrolizumab and Imatinib mesylate — In Phase Ib study:
  Level 1: Imatinib mesylate 200mg QD + Pembrolizumab 200mg Q3W, Level 2: Imatinib mesylate 400mg QD + Pembrolizumab 200mg Q3W
Drug: Pembrolizumab and Imatinib mesylate — In Phase II study, eligible patients receive the dose determined in phase Ib cohort.

SUMMARY:
This is an open-labelled single arm trial of pembrolizumab and imatinib mesylate in subjects with unresectable or metastatic KIT-mutant melanoma that are refractory to standard therapy. The phase Ib and II study will be conducted to evaluate the safety, tolerability and response rate data of this combination therapy. KIT-mutant tumors will be confirmed in previously biopsied tumors. This analysis will be done by next-generation sequencing.

DETAILED DESCRIPTION:
This trial is conducted as "Advanced medicine" authorized by the Ministry of Health, Labor, and Welfare (MHLW) in Japan, and in in conformance with Clinical Trial Act.

PIb study is a dose-escalation study comprising two dose levels of imatinib mesylate with fixed dose of pembrolizumab to evaluate safety and tolerability and identify maximum tolerated dose/administered, and determine recommended phase 2 dose (RP2D).

In PII study, a Simon's minimax two-stage design is employed.The treatment period with the combination therapy of both studies will continue every 21 days for up to 33 cycles (approximately 2 years) as long as subjects are receiving benefit from treatment and have not had disease progression or met any criteria for study withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* 1. Be male or female subjects, age 20 years or older on day of signing consent.

  2. Have histologically confirmed melanoma.

  3. Have unresectable or metastatic melanoma with KIT mutations detected by next-generation sequencing which was performed at clinical laboratories accredited by international standards such as CLIA and CAP certification.

  4. Have progressed on treatment with an anti-PD-1/L1 mAb administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression is defined by meeting all of the following criteria:
  1. Received at least 2 doses of an approved anti-PD-1/L1 mAb.
  2. Has demonstrated disease progression after PD-1/L1 as defined by RECIST 1.1. The initial evidence of disease progression is to be confirmed by second assessment no less than 4 weeks from the date of the first documented progressive disease, in the absence of rapid clinical progression. This determination is made by the investigator. Once progressive disease is confirmed, the initial date of progressive disease documentation will be considered the date of disease progression.
  3. Progressive disease has been documented within 12 weeks from the last dose of anti-PD-1/L1 mAb or during the treatment. In adjuvant therapy, progressive disease has been documented within 6 months from the last dose of anti-PD-1/L1 mAb or during the treatment.

     5. Have no prior treatment with KIT inhibitors.

     6. Have completed previous therapies 21 days prior to enrollment on study.

     7. Have the presence of at least one measurable lesion by CT or MRI per RECIST 1.1 criteria as determined by the local site investigator/radiology assessment within 14-days prior to enrollment on study.

     8. Have an Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.

     9. Have life expectancy of greater than 90 days.

     10. Have known no active central nervous system (CNS) metastases. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 28 days before enrollment on study and any neurologic symptoms).

     11. If female of childbearing potential, must be willing to use an adequate method of contraception and agree not to breastfeed for the course of the study through 120 days after the last dose of study medication. If male of childbearing potential, must agree to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication.

     12. Have laboratory parameters within Protocol-defined range. The screening laboratory tests below must be ≤14 days before enrollment on study.

  <!-- -->

  1. White blood cell count ≥ 2,000/mm^3 and absolute neutrophil count ≥1,500/mm^3.
  2. Platelets ≥ 100,000/mm^3.
  3. Hemoglobin ≥ 9 g/dL.
  4. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 150 IU/L.
  5. Bilirubin ≤ 2.0 mg/dl.
  6. Serum creatinine ≤ 1.5 mg/dl. 13. Be willing and able to review, understand and provide written consent before starting therapy.

     Exclusion Criteria:
* 1. Be seropositive for hepatitis B antigen, or hepatitis C antibody. Even if negative for HBs antigen, subjects who are positive for HBs antibody or HBc antibody and amount of HBV-DNA exceed detection sensitivity are excluded from the study.

  2. Has known history of human immunodeficiency virus（HIV) (HIV 1/2 antibodies).

  3. Has a history of (no-infectious) pneumonitis that required steroids.

  4. Has ongoing or active infections, symptomatic heart failure, unstable angina pectoris, cardiac arrhythmias, interstitial pneumonia, pneumonitis, or psychiatric disorders that would interfere with cooperation with the requirements of the study.

  5. Has known superior vena cava syndrome, pericardial effusion, pleural effusion, or ascites of grade 3 or higher.

  6. Has presence of a gastrointestinal condition that may affect drug absorption.

  7. Receiving or necessary to continue administering CYP3A4 inhibitors or drugs metabolized by CYP3A4.

  8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include cancers that have not recurred for at least 3 years before enrollment on study and early stage cancers (carcinoma in situ or stage 1) treated with curative intent, basal cell carcinoma of the skin, or superficial bladder cancer that has undergone potentially curative therapy.

  9. Has an active autoimmune disease that has required systemic treatment in past 2 years.

  10. Has history of organ transplantation including hematopoietic stem cell transplantation.

  11. Receiving chronic systemic steroid therapy. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

  12. Pregnant women and breastfeeding woman.

  13. Has received live vaccine within 30 days before the first dose of study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.

  14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Objective in phase Ib study | at 6 weeks
  Dose Limiting Toxicities (DLT) rates of pembrolizumab and imatinib mesylate combination therapy
Objective in phase II study | at 12 weeks
  Objective response rate (ORR) of treatment with recommended dose of imatinib mesylate with fixed dose of pembrolizumab according to RECIST version 1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of registration until the date of first documented disease progression or date of death from any cause, whichever came first, assessed up to 60 months.
Overall survival (OS) | From date of registration until the date of to death from any cause, assessed up to 60 months.
Best overall response (BOR) | From date of initiation of treatment until the date of the end of treatment. The maximum period for treatment is 2 years.
  BOR is defined from the overall efficacy determined by the end of this trial according to RECIST 1.1
Incidence of adverse events (AEs) graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. | Be followed up to 30 days after the cessation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Takeru Funakoshi, MD, Principal Investigator — Keio University
Locations (1):
- Keio University Hospital, Shinjuku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hirai I, Tanese K, Fukuda K, Fusumae T, Nakamura Y, Sato Y, Amagai M, Funakoshi T. Imatinib mesylate in combination with pembrolizumab in patients with advanced KIT-mutant melanoma following progression on standard therapy: A phase I/II trial and study protocol. Medicine (Baltimore). 2021 Dec 10;100(49):e27832. doi: 10.1097/MD.0000000000027832. PMID 34889232